CLINICAL TRIAL: NCT05862454
Title: Magnesium Injection Ensures Analgesia and Steroid Avoidance During Vaccination, Viremia or Immunocompromise
Brief Title: Magnesium Injection Ensures Steroid Avoidance During Vaccine, Viremia or Immunocompromise
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2022 Mg Steroid Avoid
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Steroid Metabolism Disorder
Keywords: Magnesium; Steroid avoidance
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Cohort of adult chronic pain patients, undergoing interventional injection therapy for pain management at a Canadian pain clinic
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Magnesium — Magnesium injection therapy
  Other Names: Magnesium injection

SUMMARY:
Steroid injections are used for interventional pain management. However, their side-effect of immunosuppression may increase the risk of infections. Magnesium is an alternative anti-nociceptive injection that may be used instead of steroids.

Prospective observational study of patients who received magnesium injection for interventional pain therapy, instead of steroid injection. Post-injection data collection includes numerical rating pain score, and sleep quality score. Pain is measured using the numeric pain rating scale. Sleep score is measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points is considered significant.

DETAILED DESCRIPTION:
Corticosteroid injections are used for interventional pain management. The immunosuppression effect of steroid injection may increase the risk of infections. Magnesium is an alternative anti-nociceptive agent that may be used for interventional pain injection therapy, instead of steroids.

Prospective observational clinical study of pain clinic patients who received magnesium injection for interventional pain therapy, instead of steroid injection. Post-injection data collection includes numerical rating pain score, and sleep quality score. Pain is measured using the numeric pain rating scale. Sleep score is measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points is considered significant. Data analyzed with IBM® SPSS® Statistics 25 (IBM Corp, Armonk, NY); using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* previous interventional injection therapy
* consent for interventional injection therapy
* good treatment compliance
* regular sleep diary
* regular pain diary
* informed consent for diary review
* consent for clinical record quality assurance review

Exclusion Criteria:

* organ insufficiency
* cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* unreliable diary
* poor treatment compliance
* previous adverse/allergic reactions to magnesium

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of consecutive adult patients, undergoing interventional injection therapy for pain management at a Canadian pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 12 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

SECONDARY OUTCOMES:
Sleep quality score, objective measurement using the validated Likert sleep scale | 12 weeks
  Sleep quality score, using the Likert sleep scale of 0 to 10, low scores indicate poor sleep, high scores indicate better sleep

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada